CLINICAL TRIAL: NCT02178982
Title: Standard Treatment Compliance of Participants, Effectiveness and Prognosis in Acute Respiratory Distress Syndrome
Acronym: APT
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Zhongda Hospital, Southeast University, China
Other Study IDs: ARDS protocol treatments
Record Dates: First submitted 2014-06-10; First posted 2014-07-01 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: mechanical ventilation; ARDS; Ventilator strategy; outcome
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- standard treatments of ARDS
- protocol treatment of ARDS

SUMMARY:
The Acute Respiratory Distress Syndrome (ARDS) is one of common clinical critically diseases. In the United States, the incidence of ARDS reaches 31%, which is one of the main causes of death in patients. There is no unified treatment process for ARDS currently and the treatment measures are not yet standardized, so the standardization of ARDS treatment processes is needed to reduce mortality in patients. Following the evidence-based medicine principles and six-step treatment standards of ARDS, this study uses the method of multi-center randomized controlled clinical trials to evaluate the standardized treatment process of ARDS, which provides the basis for the standardized treatment of ARDS.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* admitted to the ICU
* according to the diagnostic criteria of ARDS Berlin definition，admit patients with severe ARDS

Exclusion Criteria:

* age <18 years old
* be expected to die within 24 hours
* end-stage malignancies
* be participating in other studies, which may affect the results of this study
* DNI (do not intubation) and DNR (do not recovery) patients
* family members do not agree to sign an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of medical staff who comply the protocol treatment | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China